CLINICAL TRIAL: NCT03154697
Title: Development of Clinical Database of Individuals With Smith-Magenis Syndrome
Brief Title: Development of Clinical Database of Individuals With Smith-Magenis Syndrome and Sleep Disturbances
Status: Recruiting | Type: Observational
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00015678
Record Dates: First submitted 2017-03-16; First posted 2017-05-16 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2018-10

CONDITIONS: Sleep Disturbances in Smith-Magenis Syndrome
MeSH Terms: interventions — Spermine Synthase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection of sleep disturbances in individuals with SMS — Data related to Smith-Magenis syndrome and sleep disturbances are collected through a web or phone survey

SUMMARY:
This database will be used to better understand the sleep problems of people with SMS. This clinical database will be a part of a larger Smith-Magenis Patient Registry used to create an awareness campaign around SMS and the sleep disturbances that are characteristic of the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian of individual with Smith-Magenis Syndrome

Exclusion Criteria:

* Not legal guardian of individual with SMS

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with SMS
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of individuals with Smith- Magenis syndrome | 5 years

SECONDARY OUTCOMES:
Sleep Disturbances | Up to 100 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Pharmaceuticals, Washington D.C., District of Columbia, United States